CLINICAL TRIAL: NCT06508450
Title: Adapting and Testing A Mental Health Services Engagement Program for Racial and Ethnic Minority Young Adults
Brief Title: A Mental Health Services Engagement Program for Racial and Ethnic Minority Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: K23MH132814 (NIH)
Record Dates: First submitted 2024-07-08; First posted 2024-07-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-12

CONDITIONS: Psychosis; Bipolar and Related Disorders; Depressive Disorder
MeSH Terms: conditions — Psychotic Disorders; Bipolar and Related Disorders; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Just Do You (Active Comparator): Just Do You Core Intervention
  Interventions: Behavioral: Just Do You
- Just Do You-A (Experimental): Just Do You plus Component A
  Interventions: Behavioral: Just Do You; Behavioral: Component A
- Just Do You-B (Experimental): Just Do You plus Component B
  Interventions: Behavioral: Just Do You; Behavioral: Component B
- Just Do You-C (Experimental): Just Do You plus Component C
  Interventions: Behavioral: Just Do You; Behavioral: Component C
- Just Do You-AB (Experimental): Just Do You plus Components A and B
  Interventions: Behavioral: Just Do You; Behavioral: Component A; Behavioral: Component B
- Just Do You-AC (Experimental): Just Do You plus Components A and C
  Interventions: Behavioral: Just Do You; Behavioral: Component A; Behavioral: Component C
- Just Do You-CB (Experimental): Just Do You plus Components C and B
  Interventions: Behavioral: Just Do You; Behavioral: Component B; Behavioral: Component C
- Just Do You-ABC (Experimental): Just Do You plus Components A B and C
  Interventions: Behavioral: Just Do You; Behavioral: Component A; Behavioral: Component B; Behavioral: Component C

INTERVENTIONS:
Behavioral: Just Do You — Just Do You Core Intervention utilizes creative arts and a provider team of a licensed clinician and professional peer to increase young adult engagement in adult outpatient mental health programs. Content addresses recovery, advantages of using mental health services, working with providers, stigma, and mental health literacy.
Behavioral: Component A — Content addresses participant cultural identities and how they may be barriers and facilitators to on-going engagement with services.
  Arms: Just Do You-A; Just Do You-AB; Just Do You-ABC; Just Do You-AC
Behavioral: Component B — Content addresses identity-based motivations for on-going engagement with services and hope for the future.
  Arms: Just Do You-AB; Just Do You-ABC; Just Do You-B; Just Do You-CB
Behavioral: Component C — Content addresses community and environmental barriers and facilitators to on-going engagement with services and self-efficacy.
  Arms: Just Do You-ABC; Just Do You-AC; Just Do You-C; Just Do You-CB

SUMMARY:
Researchers aim to test a brief culturally-responsive young adult orientation program for community mental health services. They will conduct a 24-month randomized trial with 80 young adults from racial and ethnic minority groups in a community-based mental health clinic.

DETAILED DESCRIPTION:
The study objective is to assess the feasibility and acceptability of three new culturally-responsive components added to the brief young adult engagement intervention called Just Do You. The new components incorporate techniques from the DSM-5 Cultural Formulation Interview (CFI) and creative arts therapy to increase culturally-responsive content in Just Do You, which demonstrated evidence of keeping young adults connected to their treatment in a prior trial. Components are designed to elicit relevant cultural characteristics, experiences, and perspectives of diverse young adults enrolled in psychiatric rehabilitation as part of the Just Do You orientation program. The investigators will examine whether the new culturally-responsive components improve engagement in mental health services and increase service utilization.

A total of 80 young adults enrolled in an outpatient psychiatric rehabilitation program in New York will be recruited over 24 months to take part in a randomized full factorial pilot trial. Participants will be given a baseline assessment and randomly assigned to one of eight combinations of intervention components. Just Do You will be delivered first to all participants, with the assigned combination of new components to follow. The intervention will be delivered at the psychiatric rehabilitation program and will last up to five weeks for each participant, depending on the experimental condition. Outcome measures will be assessed at baseline, post-intervention, and 3-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-34
* From groups other than non-Hispanic White
* Enrolled in services at the partnering clinic site

Exclusion Criteria:

* Cognitive impairments (i.e., young adult cannot understand consent process)
* Unable to comprehend and speak English

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Participant acceptability questionnaire | Immediately after the intervention
  Self-report measure for assessing intervention acceptability from the perspectives of intervention recipients. Based on the theoretical framework of acceptability. Items are scored from 1 to 5. Possible total scores range from 9 to 45, with higher scores indicating greater acceptability.
Qualitative interviews | Immediately after the intervention
  Interviews with participants to assess acceptability of Components A, B, and C
Intervention adherence | Baseline through study completion, an average of 2 years; repeated measure to assess change through study completion
  Provider reported rate of intervention components completed by participants.

SECONDARY OUTCOMES:
Service utilization | Assessed 3 months after baseline
  Provider reported service utilization. Total number of contacts between participant and service providers starting 1 month before baseline though 3-month follow up to assess change in participant engagement.
Client Engagement in Child Protective Services Scale | Assessed immediately after the intervention and 3 months after baseline
  This scale is altered to measure young adult engagement in mental health services. The scale includes 8 questions and responses will be summed. The range for the scale is 8 to 40, with higher scores indicating higher levels of engagement.

CONTACTS AND LOCATIONS:
Locations (1):
- The Jewish Board, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moore KL, Rodwin AH, Gwadz M, Chang DF, Collins LM, Munson MR. A Brief Engagement Intervention Adapted for Racial and Ethnic Minority Young Adults in Mental Health Services: Protocol for a Pilot Optimization Trial. JMIR Res Protoc. 2025 Jun 17;14:e68885. doi: 10.2196/68885. PMID 40527500